CLINICAL TRIAL: NCT02671175
Title: Malaria Chemoprevention With Monthly Treatment With Dihydroartemisinin-piperaquine for the Post-discharge Management of Severe Anaemia in Children Aged Less Than 5 Years in Uganda and Kenya: A Two-arm Randomised Placebo Controlled Trial
Brief Title: Post-discharge Malaria Chemoprevention(PMC) Study
Acronym: PMC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: The Research Council of Norway (Other); Kenya Medical Research Institute (Other); Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 14.034; 2965 (Other: Kenya Medical Research Institute); 2015-125 (Other: Uganda REC); 2014/1911 (Other: Norway REC)
Record Dates: First submitted 2016-01-28; First posted 2016-02-02 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Malaria; Severe Anemia
MeSH Terms: conditions — Malaria; Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dihydroartemisinin-piperaquine (Active Comparator): dihydroartemisinin-piperaquine (3-day treatment courses, given 2, 6, and 10 weeks after enrollment)
  Interventions: Drug: dihydroartemisinin-piperaquine
- dihydroartemisinin-piperaquine Placebo (Placebo Comparator): Placebo comparator (matching tablets containing no active ingredients)
  Interventions: Drug: dihydroartemisinin-piperaquine placebo

INTERVENTIONS:
Drug: dihydroartemisinin-piperaquine — Children in both arms will receive standard in-hospital care for severe anaemia (blood transfusion, often combined with quinine or artesunate IV/IM). All children will then receive a 3-day course of AL (whether they initially had malaria or not), which will be started in-hospital as soon as they are able to take oral medication, and will be completed at home after discharge. At 2 weeks after enrolment surviving children will be randomized to receive either a standard 3-day courses of dihydroartemisinin-piperaquine (Eurartesim®, Sigma Tau, Italy) or an identical placebo regimen at 2, 6 and 10 weeks after enrolment.
  Other Names: Eurartesim
  Arms: dihydroartemisinin-piperaquine
Drug: dihydroartemisinin-piperaquine placebo — Children will receive standard in-hospital care for severe anaemia (blood transfusion, often combined with quinine or artesunate IV/IM). All children will then receive a 3-day course of AL (whether they initially had malaria or not), which will be started in-hospital as soon as they are able to take oral medication, and will be completed at home after discharge. At 2 weeks after enrolment surviving children will be randomized to receive either a standard 3-day courses of dihydroartemisinin-piperaquine (Eurartesim®, Sigma Tau, Italy) or an identical placebo regimen at 2, 6 and 10 weeks after enrolment.
  Other Names: Eurartesim placebo
  Arms: dihydroartemisinin-piperaquine Placebo

SUMMARY:
This study evaluates the efficacy and safety of 3 months of malaria chemoprevention post-discharge using dihydroartemisinin piperaquine (DHA-P) in children under 5 years of age admitted with severe anemia. One half will receive monthly DHA-P and the other half placebo.

DETAILED DESCRIPTION:
Children hospitalized with severe anemia in Africa are at high risk of readmission or death within 6 months after discharge. No strategy specifically addresses this post-discharge period. In Malawi, 3 months of post-discharge malaria chemoprevention with monthly 3-day treatment courses of artemether-lumefantrine (AL) in children with severe malarial anemia prevented 31% of deaths and readmissions. This study is a confirmatory efficacy trial in Kenya and Uganda to determine the efficacy and safety of malaria chemoprevention post-discharge. We hypothesize that an additional three months of malaria chemoprevention with monthly 3-day treatment courses with DHA-piperaquine (each providing about 4 weeks of post-treatment prophylaxis) provided during the post-discharge period to children recently admitted with severe anemia is superior to reduce all-cause readmission and mortality rates by 6 months compared with 2 weeks of post-treatment prophylaxis provided by the single course of oral AL when given as part of the standard in-hospital care around the time of discharge.

ELIGIBILITY:
Inclusion Criteria:

* Pre-study screening

  1. Haemoglobin <5.0 g/dl or PCV < 15%, or requirement for blood transfusion for other clinical reasons on or during admission to the hospital
  2. Aged less than 59.5 months
  3. Body weight >5 kg
  4. Resident in catchment area Enrolment in study(t=0)

  <!-- -->

  1. Fulfilled the pre-study screening eligibility criteria
  2. Aged < 59.5 months
  3. Clinically stable, able to take oral medication
  4. Subject completed blood transfusion(s) or became clinically stable without transfusion
  5. Able to feed (for breastfeeding children) or eat (for older children)
  6. Absence of know cardiac problems
  7. Provision of informed consent by parent or guardian Randomisation (t=2 weeks)

  <!-- -->

  1. Fulfilled enrolment eligibility criteria and was enrolled during recent admission
  2. Aged <60 months
  3. Still clinically stable, able to take to oral medication, able to feed (for breastfeeding children) or eat (for older children) and able to sit unaided (for older children who were already able to do so prior to hospitalisation)

Exclusion Criteria:

* Pre-study screening

  1. Recognised specific other cause of severe anaemia (e.g. trauma, haematological malignancy, known bleeding disorder)
  2. Known sickle cell disease
  3. Anticipated to reach the 5th birthday (60 months of age) within 2 weeks from enrolment (i.e. prior to randomization)
  4. Child will reside for more than 25%of the 6 months study period (i.e. 6 weeks or more) outside of catchment area Enrolment in study (t=0)

  <!-- -->

  1. Previous enrolment in the present study
  2. Known hypersensitivity to study drug
  3. Sickle cell disease
  4. Use or known need at the time of enrolment for concomitant prohibited medication during the 14 weeks PMC treatment period.
  5. Ongoing or planned participation in another clinical trial involving ongoing or scheduled treatment with prohibited medicinal products or active follow-up during the course of the study (6 months from enrolment)
  6. A known need at the time of enrolment for scheduled surgery during the subsequent course of the study (6 months from enrolment)
  7. Suspected non-compliance with the follow-up schedule
  8. Know heart conditions, or family history of congenital prolongation of the QTc interval.
  9. Taking medicinal products that are known to prolong the QTc interval Randomisation (t=2 weeks)

  <!-- -->

  1. Used dihydroartemisinin since enrolment
  2. Use or known need at the time of randomisation for concomitant prohibited medication during the 14 weeks PMC treatment period.
  3. Enrolled, or known agreement to enrol into another clinical trial involving ongoing or scheduled treatment with medicinal products during the course of the study (6 months from enrolment)
  4. A known need at the time of randomisation for scheduled surgery during the subsequent course of the study (6 months from enrolment)
  5. Suspected non-compliance with the follow-up schedule
  6. Withdrawal of consent since enrolment

Max Age: 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1049 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
All-cause deaths or all-cause re-admissions by 26 weeks from randomization (composite primary outcome). | 6 months
  Primary outcome

SECONDARY OUTCOMES:
Readmission due to severe malaria (defined as any treatment with parenteral quinine or artesunate, or presence of severe anaemia and treatment with oral antimalarials) by 26 weeks from randomization | 26 weeks from randomization
All-cause readmission by 26 weeks from randomization | 26 weeks from randomization
Readmissions due to severe anaemia (defined as Haemoglobin (Hb) <5g/dL or packed-cell volume (PCV) <15% or requirement for blood transfusion based on other clinical indication)by 26 weeks from randomization | 26 weeks from randomization
Readmission due to severe malarial anaemia (severe anaemia plus parenteral or oral antimalarial treatment)by 26 weeks from randomization | 26 from randomization
Readmission due to severe anaemia or severe malaria (composite outcome)by 26 weeks from randomization | 26 weeks from randomization
All-cause mortality by 26 weeks from randomization | 26 weeks from randomization
Clinic visits because of smear of rapid diagnostic test (RDT) confirmed non-severe malaria by 26 weeks from randomization | 26 weeks from randomization
Readmission due to severe malaria-specific anaemia (severe anaemia plus parenteral or oral antimalarial treatment and parasite density >5000/microlitre) by 26 weeks from randomization | 26 weeks from randomization
Readmission due to severe disease other than severe anaemia and severe malaria by 26 weeks from randomization | 26 weeks from randomization
Non-severe all-cause sick-child clinic visits by 26 weeks from randomization | 26 weeks from randomization
Non-malaria sick child clinic visits by 26 weeks from randomization | 26 weeks from randomization
Malaria infection at 6 month | 6 month
Hb at 6 months | 6 months
Any anaemia (Hb<11 g/dL), mild anaemia (Hb 8.0-10.99 g/dl) moderate anaemia (Hb 5.0-7.99 g/dL) and severe anaemia (Hb<5 g/dL) at 6 months | 6 months
Weight-for-age, height-for-age, and height-for-weight Z-scores, standard deviation (SD) scores of reference population) at 6 months | 6 months
Serious adverse events, excluding primary and secondary efficacy outcomes, by 26 weeks from randomization | 26 weeks from randomization
Serious adverse events within 7 days after the start of each course of PMC, excluding primary and secondary efficacy outcomes. | 26 weeks from randomization
Adverse events by 26 weeks from randomization | 26 weeks from randomization
Adverse events within 7 days after start of each course of PMC. | 7 days post drug administration
Corrected QT interval (QTc) prolongation measured by electro cardio gram (ECG)4-6 hours after 3rd dose of each course | 4-6 hours after 3rd dose of each course
Patients costs of receiving the intervention | 26 weeks after randomization
Patients costs related to treatment of the primary disease, readmission or death | 26 weeks after randomization
The costs of the health care system of providing the intervention | 26 weeks after randomization
The costs of the health system of treating the primary disease and anaemia, as well as treatment of readmissions or costs related to fatalities | 26 weeks after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Dr Titus K Kwambai, MSc, Principal Investigator — Liverpool School of Tropical Medicine; Dr Simon K Kariuki, PhD, Principal Investigator — Kenya Medical Research Institute; Dr Richard IDRO, PhD, Principal Investigator — Makerere University; Dr Robert Opoka, M.Med, Principal Investigator — Makerere University
Locations (9):
- Kenya (4):
  - Homa Bay County Referral Hospital, Homa Bay, Homa Bay County
  - Migori County Referral Hospital, Migori, Migori County
  - Siaya County Referral Hospital, Siaya, Siaya County
  - Jaramogi Oginga Odinga Teaching and Referral Hospital, Kisumu
- Uganda (5):
  - Hoima Regional Referral Hospital, Hoima
  - Jinja Regional Referral Hospital, Jinja
  - Kamuli Mission Hospital, Kamuli
  - Masaka Regional Referral Hospital, Masaka
  - Mubende Regional Referral Hospital:, Mubende

IPD SHARING:
Plan to Share IPD: Yes
All individual-participant data collected during this trial will be stored in a public data repository after de-identification. Data and documents, including the study protocol, and the statistical analysis plan, will be made available and access to data provided when a proposal has been approved by the investigators, after consideration of overlap between the proposal and any ongoing efforts. Data will be available beginning at three months after publication of this Article.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 months after publication of this Article
Access Criteria: Proposals should be directed to feiko.terkuile@lstmed.ac.uk and Bjarne.Robberstad@uib.no; to gain access, data requesters will need to sign a data access agreement, and the de-identified database will be transferred electronically

REFERENCES:
- [Derived] Kwambai TK, Dhabangi A, Idro R, Opoka R, Watson V, Kariuki S, Kuya NA, Onyango ED, Otieno K, Samuels AM, Desai MR, Boele van Hensbroek M, Wang D, John CC, Robberstad B, Phiri KS, Ter Kuile FO. Malaria Chemoprevention in the Postdischarge Management of Severe Anemia. N Engl J Med. 2020 Dec 3;383(23):2242-2254. doi: 10.1056/NEJMoa2002820. PMID 33264546
- [Derived] Kwambai TK, Dhabangi A, Idro R, Opoka R, Kariuki S, Samuels AM, Desai M, van Hensbroek MB, John CC, Robberstad B, Wang D, Phiri K, Ter Kuile FO. Malaria chemoprevention with monthly dihydroartemisinin-piperaquine for the post-discharge management of severe anaemia in children aged less than 5 years in Uganda and Kenya: study protocol for a multi-centre, two-arm, randomised, placebo-controlled, superiority trial. Trials. 2018 Nov 6;19(1):610. doi: 10.1186/s13063-018-2972-1. PMID 30400934